CLINICAL TRIAL: NCT00059423
Title: Natural History and Molecular Characterization of Benign Ethnic Neutropenia in Individuals of African Descent
Brief Title: Natural History Study for BEN
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030168; 03-H-0168
Record Dates: First submitted 2003-04-25; First posted 2003-04-25 (Estimated); Last update posted 2024-03-22 (Actual); Status verified 2020-06

CONDITIONS: Neutropenia; Agranulocytosis; Hematologic Diseases; Leukocyte Disorders; Leukopenia
Keywords: Leukapheresis; G-CSF; Dexamethasone; mRNA; Benign Ethnic Neutropenia; BEN; Healthy Volunteer; HV
MeSH Terms: conditions — Neutropenia; Agranulocytosis; Hematologic Diseases; Leukocyte Disorders; Leukopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Individuals of African descent with benign ethnic neutropenia (BEN) at baseline
- 2: Individuals of African descent without benign ethnic neutropenia (BEN) at baseline

SUMMARY:
In recent decades, hematologists have noticed that persons of African descent sometimes have lower white blood cell counts of a certain type, called granulocytes. These cells help to fight infections. The lower number of granulocytes in this situation does not appear to lead to more infections, and these individuals do not have any symptoms. This condition is called benign ethnic neutropenia (BEN), and is observed in a small percentage of individuals of African descent. This study will investigate the condition by studying people with and without BEN.

The goals of this study are to:

1. identify individuals of African descent with BEN.
2. determine the effects of two drugs, G-CSF and dexamethasone, on granulocyte production and movement.
3. determine whether there are differences in those with and without BEN in the way genes are stimulated after the administration of G-CSF and dexamethasone.

Study participants will be asked to interview with the research team, undergo physical exams, donate a blood sample, and receive G-CSF by injection, followed by dexamethasone (orally) about three weeks later. They also will be required to undergo apheresis three times, a procedure in which blood is drawn from a donor and separated into its components. Some components are retained for research analyses, such as granulocytes, and small amount of blood; the remainder is returned by transfusion to the donor. This procedure will be required of participants before they receive G-CSF, the day after they receive G-CSF, and the day after they receive dexamethasone. Gene messages (mRNA will be isolated from granulocytes, and analyzed to better understand granulocyte growth and movement.

DETAILED DESCRIPTION:
Benign ethnic neutropenia (BEN) is defined by peripheral blood absolute neutrophil count less than 1.5 x 10 (9) per liter without an increase in infections. This condition has been described in individuals of African descent. Although these individuals have normal myeloid maturation on bone marrow examinations, they appear to release fewer neutrophils into the circulation when stimulated by hydrocortisone, compared to normal controls. This suggests that there may be differences in the regulation of neutrophil release or trafficking. In the past decade, granulocyte-colony stimulating factor (G-CSF) has been widely used in a variety of clinical settings, from patients with chemotherapy-induced neutropenia to normal volunteers for peripheral blood stem cell collection. G-CSF, however, has not been used in individuals with BEN. Furthermore, gene expression in neutrophil proliferation and trafficking has not been studied in these individuals. The purpose of this study are to (1) identify individuals with BEN; (2) follow the natural history of BEN; (3) determine if there is a familial inheritance pattern; (4) characterize and compare neutrophil response to dexamethasone and G-CSF; (5) compare the pattern of neutrophil gene expression by microarray analyses; and (6) determine if mutations are present at the DNA level to account for gene expression pattern differences in individuals of African descent with and without BEN at baseline, post dexamethasone, and post G-CSF stimulation.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Individuals of African descent of age 5 or greater
* Normal renal function: creatinine <1.5 mg/dL and proteinuria <1+
* Normal liver function: bilirubin <1.5 mg/dL and transaminases within normal limits
* For control subjects: WBC within normal range (3,300-9,600/mm3), granulocytes/neutrophils greater than or equal to 2,000/mm3, platelets >150,000/mm3, hemoglobin > 11.5g/dL and normal MCV
* For benign ethnic neutropenic subjects: two blood counts, at least 1 month apart, with granulocytes/neutrophils <1,500/mm3, platelet >150,000/mm3, hemoglobin >12.5g/dL, and normal MCV. We will also follow subjects whose neutrophil counts are between 1500 and 2000/mm3 in a separate cohort periodically (e.g. once every 1-2 years) to see if their blood counts behave more like BEN or normal subjects.
* Female volunteers of childbearing age should not be pregnant
* Meets NIH Department of Transfusion Medicine (DTM) eligibility criteria for blood component donation for in vitro research uses (negative serologic tests for syphilis, hepatitis B and C, HIV, and HTLV-1)
* Ability to give informed consent to participate in the protocol

EXCLUSION CRITERIA:

* Any underlying hematologic disorder including anemia, and sickle cell disease. Subjects with thalassemia or sickle cell trait are not excluded.
* Current use of corticosteroids, e.g. prednisone, dexamethasone, or hydrocortisone. Corticosteroids must be discontinued at least one month prior
* Active or chronic viral, bacterial, fungal, or parasitic infection. Any antibiotic use should be discontinued at least one month prior
* History of autoimmune disease, such as rheumatoid arthritis or systemic lupus erythematosus, or positive anti-nuclear antibody (ANA ELISA) of 3 E.U. (ELISA units) or greater.
* Low B12 or folate levels, or abnormal thyroid function tests
* History of cancer or chemotherapy, except squamous carcinoma of the skin and cervical carcinoma in situ
* Pregnant woman or positive urine pregnancy test
* History of clinically significant cardiovascular disease (cardiology consultation may be obtained when clinically indicated)
* Any positive serum screening test as listed below
* Allergy to G-CSF or bacterial E. coli products
* Active pulmonary disease or a pulse-ox level of less than 95% on screening exam

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Since BEN is a condition of individuals of African descent, volunteer recruitment will be focused in this ethnic population. Accrual for BEN subjects will be based on entry criteria, and not on gender or age (in those 5 years or greater). The minimum age is 5 years because these older children would have larger veins and would be more likely to cooperate with blood draws. Subjects without BEN will be selected to match age and gender of BEN subjects to minimize the differential effects of age and gender to the responses to G-CSF and dexamethasone and in microarray analyses.
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2003-06-03 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Serial blood counts in BEN | Ongoing
  In our study, we hope to further elucidate the etiology of BEN in research subjects by isolating granulocyte mRNA after G-CSF and dexamethasone stimulation, applying microarray analyses to screen for gene expression differences, and confirming expression pattern differences by DNA analyses. We will focus on genes that are important in the proliferation and trafficking of neutrophils,such as PRV-1, elastase, myeloblastin, transcription factor PU.1, CAAT enhancing binding protein-alpha (C /EBP), stromal derived factor-1 (SDF-1), and CXC receptor-4 (CXCR4).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew M Hsieh, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ash RC, Mendelsohn LA, Marshall ME. Hemopoietic marrow function in chronic neutropenia of blacks: cure of aplastic anemia by allogeneic marrow transplantation from a neutropenic sibling donor. Am J Hematol. 1986 Jun;22(2):205-12. doi: 10.1002/ajh.2830220212. PMID 3518419
- [Background] Haddy TB, Rana SR, Castro O. Benign ethnic neutropenia: what is a normal absolute neutrophil count? J Lab Clin Med. 1999 Jan;133(1):15-22. doi: 10.1053/lc.1999.v133.a94931. PMID 10385477
- [Background] Mason BA, Lessin L, Schechter GP. Marrow granulocyte reserves in black Americans. Hydrocortisone-induced granulocytosis in the "benign" neutropenia of the black. Am J Med. 1979 Aug;67(2):201-5. doi: 10.1016/0002-9343(79)90391-7. PMID 463924
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-H-0168.html